CLINICAL TRIAL: NCT03960658
Title: Repeated Sub-anesthetic Ketamine to Enhance Prolonged Exposure Therapy in Post-traumatic Stress Disorder: A Proof-of-concept Study
Brief Title: Ketamine and Prolonged Exposure in PTSD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paulo Shiroma, Clinical Investigator, Minneapolis Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAM-18-00333
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Results first posted 2021-03-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine and PE (Experimental): ketamine treatment followed by a standardized prolonged exposure session for the first 3 weeks; then, weekly prolonged exposure as usual.
  Interventions: Drug: ketamine-enhanced prolonged exposure

INTERVENTIONS:
Drug: ketamine-enhanced prolonged exposure — Subjects will receive a single infusion of racemic ketamine at 0.5mg/kg (ideal body weight) for 40 minutes. The next day, patients will have a standardized prolonged exposure session which lasts approximately 90 minutes. This co-jointed intervention will be repeated for 3 weeks. Then, patients will continue with therapy sessions to complete a total of 10-12 sessions.

SUMMARY:
This study aims at investigating the effectiveness of the drug, Ketamine, in combination with Prolonged Exposure (PE) therapy for people suffering from PTSD. Participation in the study includes Ketamine infusions, which occur once a week for three weeks. PE therapy sessions will be scheduled one day after each infusion, and may continue up to 12 weeks. After completely therapy, there will be two monthly follow-up assessment visits.

DETAILED DESCRIPTION:
Study location: Minneapolis VA Medical Center

The study is an open-label interventional study designed to inform and strengthen the feasibility of protocol implementation on sub-anesthetic doses of intravenous Ketamine as augmenting strategy of standardized, manually-driven Prolonged Exposure therapy in PTSD.

Timeline: Eligible individuals can expect their participation to last up to 5 months. Compensation will be given for participation per session that is attended. Potential participants will be provided with information about the study and asked a series of questions to determine if they meet basic inclusion/exclusion criteria (e.g., indicators of current PTSD). They will be informed that the treatment involves multiple infusions of sedatives at subanesthetic doses followed by PE therapy. Those interested will be scheduled for an in-person, baseline session.

Voluntary informed consent will be obtained in accordance with local IRB approvals. During the baseline, all assessments, computer tasks, and information on treatment will be explained. Participants will also undergo a urine toxicology analysis during this session. Ketamine infusions and PE therapy appointments will be scheduled within two weeks of the baseline.

The day of the infusion, patients will arrive in the morning after an overnight fast of at least 8 hours. An IV will be placed in the non-dominant arm for medication administration. Vitals will be recorded throughout the entire medication treatment. Subjects will then receive IV infusion of 0.5mg/Kg of ketamine hydrochloride solution over 40 minutes. The dose of ketamine will be calculated by ideal body weight. Any altered sensory or dissociative effects will be measured before and after each infusion. Vitals will be monitored for another hour, until all side-effects have subsided. Participants are required not to drive or use heavy machinery until the following morning.

One day after the infusion, patients will come back for study assessments and Prolonged Exposure therapy with a VA psychologist. PE is an evidence-based psychotherapy for PTSD that is based on the Emotional Processing Theory of PTSD; the four components of PE are: 1) exposure to safe situations, objects, or people that cause distress and are avoided because they are trauma reminders (in vivo exposure), 2) revisiting and processing of the trauma memory (imaginal exposure), 3) psycho-education about trauma-related symptoms, and 4) breathing retraining. Session 1 includes the presentation of treatment rationale and program overview, information gathering, and breathing retraining. Session 2 includes education about common reactions to trauma, rationale for in vivo exposure, and construction of an in vivo exposure hierarchy. The hierarchy includes safe or low-risk activities and situations that were avoided because of their association with the trauma. Throughout the treatment, participants will be assigned homework to confront items on the hierarchy in a gradual fashion, working up to the most anxiety-arousing situations. During Session 3, the rationale for confronting the trauma memory in imagination is presented and initiation of imaginal exposure and processing is conducted. In this procedure, participants will be asked to close their eyes, visualize the trauma, and recount it aloud in the present tense for 45-60 min. The memory recounting will be repeated if necessary to allow total reliving of 45-60 min. The exposure will be audiotaped; participants will be instructed to listen daily to the tape. Sessions 4-10 will be conducted in a similar fashion: therapists review homework, conduct imaginal exposure to trauma memory for 30-45 min, discuss the imaginal exposure, and assigned in vivo and imaginal exposure homework. In the final session, participants summarize learning in treatment, discuss their progress, plans, and relapse prevention.

Upon PE completion, participants are asked to come back for 2 follow-up sessions over two months. Familiar study and PTSD assessments will be administered during this time.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of chronic (minimum of three months) PTSD (Clinician-Administered PTSD Scale for DSM-5 -CAPS-5 score>33).
2. Voluntarily eligible to participate in PE.
3. Severity of PTSD symptoms defined by PCL-5>33.
4. Psychotropic medications on stable doses (no dosing adjustments/changes for ≥4 weeks; ≥6 weeks for fluoxetine) prior to prior to beginning of the study.

Exclusion Criteria:

1. Unwillingness/unable to sign informed consent.
2. Previous or current participation in trauma-exposed therapy and/or ketamine treatment.
3. Evidence of mental retardation, pervasive developmental disorder and/or moderate/severe cognitive impairment (MMSE scores ≤27).
4. Any unstable medical or non-psychiatric CNS condition.
5. Lifetime history of psychosis-related disorder, bipolar disorder I or II disorder, or any condition other than PTSD judged to be the primary presenting psychiatric diagnosis.
6. Moderate to severe traumatic brain injury (mental status change or loss of consciousness>30 min; Glasgow Coma Scale <13; post-traumatic amnesia>24hours; visible lesion on CT/MRI brain scan).
7. Active alcohol/illicit substance use disorder within 6 months of initial assessment; presence of illicit drugs by positive urine toxicology.
8. For women: pregnancy (confirmed by lab test), initiation of female hormonal treatments within 3 months of screening, or inability/ unwillingness to use a medically accepted contraceptive method during the study.
9. Imminent risk of suicidal/homicidal ideation and/or behavior with intent and/or plan

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo R Shiroma, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shiroma PR, Thuras P, Wels J, Erbes C, Kehle-Forbes S, Polusny M. A Proof-of-Concept Study of Subanesthetic Intravenous Ketamine Combined With Prolonged Exposure Therapy Among Veterans With Posttraumatic Stress Disorder. J Clin Psychiatry. 2020 Nov 10;81(6):20l13406. doi: 10.4088/JCP.20l13406. No abstract available. PMID 33176074

RESULTS

PARTICIPANT FLOW:
Groups:
- Ketamine and Prolonged Exposure: Open-label intravenous ketamine 0.5 mg/kg 24 hours prior to prolonged exposure (PE) session 1,2 and 3 followed by up to 7 additional PE sessions.
Period: Overall Study
Arm/Group | Ketamine and Prolonged Exposure
Started | 12
Completed | 10
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ketamine and Prolonged Exposure
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Post-traumatic Stress Disorder Check List DSM-5 [Mean (Standard Deviation); unit: units on a scale] | 56.3 (9.8)
Montgomery-Åsberg Depression rating Scale [Mean (Standard Deviation); unit: units on a scale] | 25.0 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Post-traumatic Stress Disorder (PTSD) Symptoms
Description: The overall severity of PTSD symptoms would be measured by the mean change in the Past Month (current) total scores on the Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (CAPS-5) from baseline to post-treatment (10 weeks). The CAPS-5 is a structured interview with higher values representing worse outcomes. The CAPS-5 total symptom severity score ranges from 0 to 80 and it is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms.
Time Frame: 10 weeks
Population: mean CAPS-5 score at 10 weeks minus mean CAPS-5 score at baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ketamine and Prolonged Exposure
Number analyzed (Participants) | 10
units on a scale | 15.3 [7.3 to 23.2]

2. Secondary Outcome: Change in Severity of Depressive Symptoms
Description: Total score on the Montgomery- Åsberg Depression Rating Scale , a semi- structured 10-item scale. Range 0-60. Higher values represent worse outcomes. The total score is obtained by summing the severity score of each item.
Time Frame: 10 weeks
Population: mean MADRS score at 10 weeks minus mean MADRS score at baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Ketamine and Prolonged Exposure
Number analyzed (Participants) | 10
units on a scale | 11.5 [6.1 to 16.9]

3. Secondary Outcome: Change in PTSD Symptoms for DSM-5
Description: The PTSD Checklist for DSM-5 (PCL5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Range from 0-80. Higher values represent worse outcomes.
Time Frame: 10 weeks
Population: mean PCL-5 score at 10 weeks minus mean PCL-5 score at baseline
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ketamine and Prolonged Exposure
Number analyzed (Participants) | 10
score on a scale | 30.8 [20.1 to 41.4]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Ketamine and Prolonged Exposure
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 3/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine and Prolonged Exposure (N=10)
nausea (Gastrointestinal disorders) | 1 (2)
high blood pressure (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT03960658/Prot_SAP_000.pdf